CLINICAL TRIAL: NCT03291340
Title: A Pilot Cross-sectional Cohort Study of Right-to-left-shunt, Cerebrovascular Reactivity, Ischemic Infarct Burden on High Resolution MRI, and Cognitive Impairment in Elderly Subjects
Brief Title: Determining the Impact of Shunting and CerebroVascular Reactivity on 7T MRI (DISCoVeR 7T MRI)
Acronym: DISCoVeR
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Steven Messe, Associate Professor of Neurology, University of Pennsylvania
Other Study IDs: 827852
Record Dates: First submitted 2017-09-15; First posted 2017-09-25 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cognitively normal elderly: TCD agitated saline right-to-left shunt study TCD cerebrovascular reactivity study
- Cognitive impaired elderly: TCD agitated saline right-to-left shunt study TCD cerebrovascular reactivity study

SUMMARY:
The purpose of this study is to use transcanial doppler (TCD) ultrasound to look for possible risk factors for ischemic brain injury. We will perform contrast TCD with agitated saline contrast to identify and contrast right-to-left shunt (RLS) and breath holding to assess cerebrovascular reactivity (CVR) in the elderly.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 60 years of age.
2. Fluent in English.
3. Part of the NACC longitudinal cohort (Protocol #: 068200) of the PMC/ADCC with consensus conference designation of cognitively normal, Mild Cognitive Impairment, or probable/possible Alzheimer's disease.
4. Has consented to participate in the ADCC high-resolution MRI sub-study.
5. NACC longitudinal visit must be within 6 months of the TCD study and brain MRI study.
6. Women: post-menopausal or surgically sterile.
7. Willing and able to complete all required study procedures.
8. Completed 6 grades of education.
9. Geriatric Depression scale less than 6 (assessed within 6 months at the NACC longitudinal visit).

Exclusion Criteria:

1. Prior clinically symptomatic ischemic or hemorrhagic stroke.
2. Inability to tolerate or contraindication to TCD study in the opinion of an investigator or treating physician.
3. Any medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Only subjects that are enrolled in the NACC longitudinal cohort (Protocol 068200) will be eligible for this study. Subjects must also agree to participate in the ADCC high-resolution MRI sub-study to be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Presence of right-to-left shunt on TCD | Baseline
Presence of cerebrovascular reactivity on TCD | Baseline

SECONDARY OUTCOMES:
Volume of ischemic injury | Baseline
Location of ischemic injury | Baseline
Presence of cognitive impairment | Baseline
Type of cognitive impairment | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No